CLINICAL TRIAL: NCT05375942
Title: Characteristics and 6-month Outcomes Among Real-World Rheumatoid Arthritis Patients Initiating Inflectra
Brief Title: This is a Retrospective Observational Study Looking at the Characteristics and Outcomes of Participants Taking Inflectra Using the CorEvitas Rheumatoid Arthritis Registry
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C1231007
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Results first posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2023-10

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- characteristics of patients newly initiated on Inflectra
  Interventions: Drug: Inflectra
- outcomes after initiating Inflectra
  Interventions: Drug: Inflectra

INTERVENTIONS:
Drug: Inflectra — 1. To describe the characteristics of patients newly initiated on Inflectra.
  Groups: characteristics of patients newly initiated on Inflectra
Drug: Inflectra — 2. To describe 6-month outcomes after initiating Inflectra, among patients who have 6 months follow-up information in the CorEvitas' RA Registry.
  Groups: outcomes after initiating Inflectra

SUMMARY:
This is a retrospective observational study looking at the characteristics and outcomes of participants taking Inflectra using the CorEvitas Rheumatoid Arthritis Registry.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age
* Have been diagnosed with RA by a rheumatologist
* Have initiated treatment with Inflectra
* Had assessment of effectiveness in patients who have at least one follow up visit.

Exclusion Criteria:

* No additional exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective analysis of an existing database of patient encounters from the CorEvitas RA Registry
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Collegeville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1231007

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of participants with Rheumatoid Arthritis (RA) who had initiated Inflectra was retrieved from the CorEvitas RA registry and observed in this retrospective observational study.
Groups:
- All Participants (Cohort 1): All participants diagnosed with RA who were Inflectra initiators in real world, who met inclusion criteria, and whose data were observed in this study.
Period: Overall Study
Arm/Group | All Participants (Cohort 1)
Started | 255
Participants With 6 Month Follow-up (Cohort 2) | 176
Completed | 255
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All eligible participants whose data was observed in this study.
Arm/Group | All Participants (Cohort 1)
Number analyzed (Participants) | 255
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Data is presented for participants evaluable in Cohort 1 and 2.
  Years
    Cohort 1 | 64.0 (12.7)
    Cohort 2: number analyzed (Participants) | 176
    Cohort 2 | 63.6 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data is presented for participants evaluable in Cohort 1 and 2.
  Participants
    Cohort 1: Female | 194
    Cohort 1: Male | 61
    Cohort 2: number analyzed (Participants) | 176
    Cohort 2: Female | 138
    Cohort 2: Male | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Data is presented for participants evaluable in Cohort 1 and 2.
  Participants
    Cohort 1: White | 192
    Cohort 1: Non-white | 62
    Cohort 1: Not reported | 1
    Cohort 2: number analyzed (Participants) | 176
    Cohort 2: White | 133
    Cohort 2: Non-white | 43
    Cohort 2: Not reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Low Disease Activity (LDA) at 6 Months After Inflectra Initiation
Description: Clinical disease activity index (CDAI) was the numerical sum of 4 outcome parameters: tender and swollen joint count based on a 28-joint assessment, participant global assessment and physician global assessment assessed on 0 to 10 millimeter (mm) visual analogue scale (VAS) where 0 mm = minimum possible pain (best) and 100 mm = maximum possible pain (worst). Total score for CDAI ranged from 0 to 76 with higher score indicating greater disease activity. Participants who achieved LDA had CDAI score less than or equal to (<=)10. Participants with moderate or high disease activity (CDAI greater than [>]10) at baseline were analyzed for this outcome measure.
Time Frame: 6 Months (from the retrospective data collected from the CorEvitas RA registry)
Population: All eligible participants who had CDAI available at baseline and at 6-months follow-up visit and CDAI measured at the 6-month follow-up visit. Here "Number of Participants Analyzed" signifies number of participants with moderate or high disease activity (CDAI>10) at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Participants With 6-Months Follow-up (Cohort 2): All participants diagnosed with RA who were Inflectra initiators in real world, who met inclusion criteria, and had CDAI available at Baseline and at 6-months follow-up visit.
Arm/Group | Participants With 6-Months Follow-up (Cohort 2)
Number analyzed (Participants) | 85
Percentage of participants | 32.9 [22.9 to 42.9]

2. Secondary Outcome: Percentage of Participants Who Achieved Clinical Remission at 6 Months After Inflectra Initiation
Description: CDAI was the numerical sum of 4 outcome parameters: tender and swollen joint count based on a 28-joint assessment, participant global assessment and physician global assessment assessed on 0 to 10 mm VAS where 0 mm = minimum possible pain (best) and 100 mm = maximum possible pain (worst). Total score for CDAI ranged from 0 to 76 with higher score indicating greater disease activity. Participants who achieved clinical remission had a CDAI score <=2.8. Participants with low, moderate or high disease activity (CDAI>2.8) at baseline were analyzed for this outcome measure.
Time Frame: 6 Months (from the retrospective data collected from the CorEvitas RA registry)
Population: All eligible participants who had CDAI available at baseline and at 6-months follow-up visit and CDAI measured at the 6-month follow-up visit. Here "Number of Participants Analyzed" signifies number of participants with moderate or high disease activity (CDAI>2.8) at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Participants With 6-Months Follow-up (Cohort 2)
Number analyzed (Participants) | 131
Percentage of Participants | 13.7 [7.8 to 19.6]

3. Secondary Outcome: Change From Baseline in CDAI at 6 Months After Inflectra Initiation
Description: CDAI was the numerical sum of 4 outcome parameters: tender and swollen joint count based on a 28-joint assessment, participant global assessment and physician global assessment assessed on 0 to 10 mm VAS where 0 mm = minimum possible pain (best) and 100 mm = maximum possible pain (worst). CDAI total score = 0 to 76, higher scores=greater affection due to disease activity. CDAI <2.8 indicated disease remission, 2.8 to <10 indicated low disease activity, 10 to <22 indicated moderate disease activity, and >=22 indicated high disease activity.
Time Frame: Baseline, 6 Months (from the retrospective data collected from the CorEvitas RA registry)
Population: All eligible participants who had CDAI available at baseline and at 6-months follow-up visit and CDAI measured at the 6-month follow-up visit.
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Participants With 6-Months Follow-up (Cohort 2)
Number analyzed (Participants) | 176
Units on scale | -1.8 (10.0)

4. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire (HAQ) at 6 Months After Inflectra Initiation
Description: HAQ: participant-reported questionnaire for the assessment of rheumatoid arthritis. It comprised of 20 questions in 8 categories of activities: dress/groom; arise; eat; grip; walk; hygiene; reach; and activities over past week. Each activity was assessed on a 4-point Likert scale from 0 to 3, where 0 = without difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score ranged from 0 to 3, where 0 = least difficulty and 3 = extreme difficulty, higher scores indicating worse functioning.
Time Frame: Baseline, 6 Months (from the retrospective data collected from the CorEvitas RA registry)
Population: All eligible participants who had CDAI available at baseline and at 6-months follow-up visit and CDAI measured at the 6-month follow-up visit. Here "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Participants With 6-Months Follow-up (Cohort 2)
Number analyzed (Participants) | 85
Units on scale | -0.0 (0.4)

5. Secondary Outcome: Change From Baseline in Participant Pain Assessment at 6 Months After Inflectra Initiation
Description: Participant pain was measured on a VAS where 0 mm = minimum possible pain (best) and 100 mm = maximum possible pain (worst).
Time Frame: Baseline, 6 Months (from the retrospective data collected from the CorEvitas RA registry)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | Participants With 6-Months Follow-up (Cohort 2)
Number analyzed (Participants) | 176
Millimeter | -0.5 (22.4)

6. Secondary Outcome: Change From Baseline in Participant Fatigue Assessment at 6 Months After Inflectra Initiation
Description: Participant fatigue was measured on a VAS, where 0 mm = no fatigue and 100 mm = worst possible fatigue.
Time Frame: Baseline, 6 Months (from the retrospective data collected from the CorEvitas RA registry)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | Participants With 6-Months Follow-up (Cohort 2)
Number analyzed (Participants) | 176
Millimeter | -1.4 (24.4)

7. Secondary Outcome: Percentage of Participants With a Modified American College of Rheumatology 20 Percent (%) (mACR20) Response at 6 Months After Inflectra Initiation
Description: mACR20 response: >= 20% improvement in tender and swollen joint count and 20% improvement in two of the following four criteria: 1) participant assessment of pain (scored from 0 mm to 100 mm, higher scores indicated worsening of pain); 2) participant global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 3) physician global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 4) self-assessed disability index of the mHAQ (scored from 0 to 3, higher scores indicated worsening of function).
Time Frame: 6 Months (from the retrospective data collected from the CorEvitas RA registry)
Population: All eligible participants who had CDAI available at baseline and at 6-months follow-up visit and CDAI measured at the 6-month follow-up visit. Here "Number of Participants Analyzed" signifies number of participants with complete information for calculation of mACR.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Participants With 6-Months Follow-up (Cohort 2)
Number analyzed (Participants) | 167
Percentage of participants | 12.6 [7.5 to 17.6]

8. Secondary Outcome: Percentage of Participants With mACR50 at 6 Months After Inflectra Initiation
Description: mACR50 response: >= 50% improvement in tender and swollen joint count and 50% improvement in two of the following four criteria: 1) participant assessment of pain (scored from 0 mm to 100 mm, higher scores indicated worsening of pain); 2) participant global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 3) physician global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 4) self-assessed disability index of the mHAQ (scored from 0 to 3, higher scores indicated worsening of function).
Time Frame: 6 Months (from the retrospective data collected from the CorEvitas RA registry)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Participants With 6-Months Follow-up (Cohort 2)
Number analyzed (Participants) | 167
Percentage of participants | 8.4 [4.2 to 12.6]

9. Secondary Outcome: Percentage of Participants With mACR70 at 6 Months After Inflectra Initiation
Description: mACR70 response: >= 70% improvement in tender and swollen joint count and 70% improvement in two of the following four criteria: 1) participant assessment of pain (scored from 0 mm to 100 mm, higher scores indicated worsening of pain); 2) participant global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 3) physician global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 4) self-assessed disability index of the mHAQ (scored from 0 to 3, higher scores indicated worsening of function).
Time Frame: 6 Months (from the retrospective data collected from the CorEvitas RA registry)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Participants With 6-Months Follow-up (Cohort 2)
Number analyzed (Participants) | 167
Percentage of participants | 4.2 [1.2 to 7.2]

ADVERSE EVENTS:
Time Frame: Not applicable for this study as safety data was not planned to be collected during the study
Description: In the study, individual participant data were not retrieved or validated, and it was not possible to link (ie, identify a potential association between) a particular product and medical event for any individual. Thus, the minimum criteria for reporting an adverse event (AE) (ie, identifiable participant, identifiable reporter, a suspect product, and event) could not be met.
Arm/Group | All Participants (Cohort 1) | Participants With 6-Months Follow-up (Cohort 2)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-07-24): https://cdn.clinicaltrials.gov/large-docs/42/NCT05375942/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-29): https://cdn.clinicaltrials.gov/large-docs/42/NCT05375942/SAP_001.pdf